CLINICAL TRIAL: NCT04271059
Title: The Effect of Platelet Bioenergetics in Traumatic Brain Injuries
Brief Title: Platelet Bioenergetics in TBI
Status: Terminated | Type: Observational
Why Stopped: Low recruitment
Sponsor: Kevin Hatton (Other)
Responsible Party: Sponsor-Investigator, Kevin Hatton, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 54012
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Brain Injuries, Traumatic
Keywords: TBI
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- TBI without polytrauma: Subjects who have experienced a severe traumatic brain injury (Glasgow Coma Scale (GCS) 3-13) within the last 12 hours, without additional polytrauma.
- TBI with polytrauma: Subjects who have experienced a severe traumatic brain injury (Glasgow Coma Scale (GCS) 3-13) and polytrauma, including major trauma to the chest, abdomen, pelvis or extremities. within the last 12 hours.
- Healthy Control: Subjects who have not experienced any TBIs within the last six months.

SUMMARY:
This is a prospective study enrolling 5 patients with a diagnosis of traumatic brain injury (TBI) without polytrauma and 5 patients with TBI with polytrauma admitted to the University of Kentucky (UK) Chandler Medical Center to evaluate differences in platelet bioenergetics in the populations. Additionally, five healthy subjects will be recruited to the control group.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is used to describe a myriad of primary and secondary brain-related injuries related to trauma. Clinically, moderate-to-severe brain injury results in early coagulopathy, with a tendency toward unanticipated bleeding, followed by delayed hypercoagulation, with a tendency toward unanticipated clot formation. Optimal platelet count, activation and function are necessary for normal coagulation. Investigators have recently developed a novel approach to measure platelet activity. This approach specifically measures platelet energy output or bioenergetics from blood samples. Preclinical (animal) studies show that platelet bioenergetic profiles are different after TBI and that they change over time. This temporal profile may be used as a biomarker that can inform diagnosis and prognosis of TBI.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have moderate to severe traumatic brain injury (Glasgow Coma Scale (GCS) 3-13) to be enrolled in the TBI or TBI with trauma groups.
* Patients enrolled in the TBI with polytrauma group must also exhibit polytrauma including concomitant traumatic brain injury, major trauma to the chest, abdomen, pelvis or extremities.
* Patients must be greater than or equal to 18 years of age and must be less than or equal to 50 years of age.
* Patients must be able to cooperate for a detailed neurologic exam.
* Patients must be consented and undergo first blood sampling within the first 12 hours (+/- 2 hours) after their traumatic brain injury to be enrolled in the TBI or TBI with trauma groups.
* Patients must be expected to survive to discharge, as assessed by their admitting neurosurgery team

Exclusion Criteria:

* For the control group only, patients who have experienced a TBI in the last 6 months.
* Diagnosis of platelet diseases or disorders, such as thrombocytopenia, thrombocytosis, or Von Willebrand disease.
* Platelet transfusion within the last six months.
* Comorbid regimen of Metformin within the last 6 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Up to fifteen (15) subjects, who are between the ages of 18-50, including both males and females, from all ethnic and racial backgrounds will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-02-13 (Actual)

PRIMARY OUTCOMES:
Change in Platelet Bioenergetics | 0-72 hours
  Change in various platelet oxygen consumption rates and extracellular acidification rate

SECONDARY OUTCOMES:
Identify platelet bioenergetic rate of healthy adults. | 24 hour.
  Identify normal platelet oxygen consumption rates and extracellular acidification rate based on patient demographics.

CONTACTS AND LOCATIONS:
Overall Officials: kevin Hatton, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No